CLINICAL TRIAL: NCT07269080
Title: STM-06: POLARIS-POlymetastic Lesion Ablative Radiotherapy With Immunotherapy Study
Acronym: STM-06
Status: Recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: University of Illinois at Chicago (Other)
Responsible Party: Principal Investigator, Ryan Nguyen, Principal Investigator, University of Illinois at Chicago
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 2025-0362
Record Dates: First submitted 2025-11-21; First posted 2025-12-08 (Actual); Last update posted 2025-12-17 (Actual); Status verified 2025-12

CONDITIONS: Advanced Solid Tumor; Metastatic Cancer
MeSH Terms: conditions — Neoplasm Metastasis

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: No

ARMS (2):
- Treatment with Radiotherapy in Participants with Stable Disease or Partial Response (Other): Participants with investigator-assessed stable disease or partial response after > 3 months of immunotherapy treatment prior to registration
  Interventions: Radiation: Ablative radiation treatment
- Treatment with Radiotherapy in Patients with Oligo-progression (Other): Participants with oligo-progression defined as having at least 3 sites of disease during their disease course, with at least 1 but up to 5 sites of progressive disease within 3 months of registration. Participants must have investigator-assessed stable disease, partial response, or complete response as prior best response to immunotherapy and have been on immunotherapy for at least 3 months prior to registration.
  Interventions: Radiation: Ablative radiation treatment

INTERVENTIONS:
Radiation: Ablative radiation treatment — Ablative radiation for all metastases should be completed within 3 weeks of the first dose of radiation. Metastases may be treated on an everyday or every other day schedule.

SUMMARY:
This is a non-randomized two-arm trial, specifically a pilot study in which patients with advanced solid tumor cancer with 3-10 metastatic lesions who are on immunotherapy will receive ablative RT to up to 10 lesions. After study intervention, participants will undergo ctDNA collection at 8 weeks after completion of ablative RT Post-treatment disease assessments, including imaging and serial ctDNA monitoring, as well as any additional treatments, will be at the discretion of the treating oncologist. Approximately 28 subjects (14 per cohort) will be enrolled. For subjects who do not complete the full planned course of RT for any reason, a final study visit should be performed approximately 30 days after the last fraction of radiation. If a subject is discontinued from the study with an ongoing adverse event or an unresolved clinically significant laboratory result, the clinical investigative team will attempt to provide follow-up until a satisfactory clinical resolution of the laboratory result or adverse event is achieved.

ELIGIBILITY:
Inclusion Criteria:

* Age ≥ 18 years of age at the time of consent
* ECOG (0, 1, or 2) within 30 days prior to registration.
* Subjects with advanced solid tumors with at least 3 but no more than 10 sites of metastatic disease, excluding the primary tumor.
* Disease site must be outside of the GI tract (including esophagus, stomach, small or large bowel, and mesenteric lymph nodes), brainstem, and skin.
* Demonstrates adequate organ function. All screening labs are to be obtained within 30 days prior to registration.
* Able to provide written informed consent and HIPAA authorization for release of personal health information via an approved UIC Institutional Review Board (IRB) informed consent form and HIPAA authorization. If a subject is unable to consent, a Legally Authorized Representative (LAR) may provide consent on their behalf.
* Women of childbearing potential must not be pregnant or breastfeeding. A negative serum or urine pregnancy test is required per institutional practice guidelines.
* As determined at the discretion of the enrolling physician or protocol designee, the ability of the subject to understand and comply with study procedures for the entire length of the study.
* Have a life expectancy of at least 3 months.
* Subjects receiving treatment for >3 months with an FDA-approved immunotherapy agent such as a PD-1 inhibitor, a PD-L1 inhibitor, a CTLA-4 inhibitor, or an LAG-3 inhibitor; either as monotherapy or in combination with another FDA-approved immunotherapy agent. Subjects may have received prior combination cytotoxic chemotherapy and immunotherapy, but must be receiving only immunotherapy for at least 30 days prior to registration.

  * Cohort A: Subjects with investigator-assessed stable disease or partial response after > 3 months of immunotherapy treatment prior to registration
  * Cohort B: Subjects with oligo-progression defined as having at least 3 sites of disease during their disease course, with at least 1 but up to 5 sites of progressive disease within 3 months of registration. Subjects must have investigator-assessed stable disease, partial response, or complete response as prior best response to immunotherapy and have been on immunotherapy for at least 3 months prior to registration.

Exclusion Criteria:

* Inability to treat all sites of disease
* >10 metastatic lesions at any point in the disease course
* History of interstitial lung disease or G3 or worse pneumonitis
* Malignant pleural effusion
* Active infection requiring IV antibiotics
* Active autoimmune disease requiring immunosuppression in the last two years from enrollment.
* Significant medical comorbidities precluding radiotherapy as determined by the treating physician.
* Use of systemic corticosteroids equivalent to prednisone ≥10 mg daily within 14 days prior to registration, or requirement for systemic corticosteroids at screening for disease control, unless used as physiologic replacement (e.g., adrenal insufficiency). Subjects who require systemic steroids ≥10 mg/day for clinical management will be ineligible.
* Substantial overlap with a previously treated radiation volume.
* For patients with liver metastases, moderate/severe liver dysfunction (Child-Pugh B or C)
* Patients with symptomatic brain metastases, a single metastasis greater than 5 cm in size, or any brain metastasis greater than 3 cm in size. Patients with total brain metastases volume exceeding 30 cc.
* Clinical or radiologic evidence of spinal cord compression.
* Metastatic disease involving the GI tract (esophagus, stomach, small or large bowel, mesenteric lymph nodes), disease in the brainstem, or skin
* Pregnant or nursing
* Any prior or concurrent malignancy whose natural history or treatment has the potential to interfere with the safety or efficacy assessment of this investigational regimen, as determined by the treating medical oncologist.
* Other major comorbidity, as determined by the study PI

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 28 (Estimated)
Dates: Start 2025-12-08 (Actual); Primary Completion 2028-01 (Estimated); Study Completion 2028-11 (Estimated)

PRIMARY OUTCOMES:
To estimate the proportion of patients with advanced tumors and polymetastatic disease on immunotherapy who achieve a molecular response (>50% ctDNA reduction) at 8 weeks following ablative radiation therapy | Baseline to 8 weeks following the end of ablative radiation therapy

SECONDARY OUTCOMES:
To evaluate 6-month and 12-month overall survival (OS) | Registration date until the off-study date, approximately 12 months after the end of radiation therapy
  Overall survival is defined as the time from the first dose to death due to any cause, incidence of serious adverse events in all groups according to CTCAE
To evaluate 6-month and 12-month progression-free survival (PFS) | Registration date until the off-study date, approximately 12 months after the end of radiation therapy
  Progression-free survival is defined as the time from the time of enrollment to disease progression or death, whichever occurs first
To evaluate overall response rate | Registration date until the off-study date, approximately 12 months after the end of radiation therapy
  Overall response rate is defined as partial response (PR) or complete response (CR) occurring at any point during treatment, as assessed by the treating physician
To evaluate all grades of treatment-related adverse events (TRAEs) | Treatment start until the off-study date, approximately 12 months after the end of radiation therapy
  Treatment related adverse events will be assessed by CTCAE version 5.

OTHER OUTCOMES:
To assess the concentration of circulating immune cells before and after concurrent radiation and immunotherapy | Baseline until 48 weeks post-radiation treatment

CONTACTS AND LOCATIONS:
Overall Officials: Ryan Nguyen, DO, Principal Investigator — University of Illinois at Chicago
Locations (1):
- University of Illinois at Chicago, Chicago, Illinois, United States